CLINICAL TRIAL: NCT00144001
Title: Appropriateness of Antiepileptic Drug Use for Older Veterans
Brief Title: Factors Associated With in Suboptimal Prescribing for Older Patients With Epilepsy
Acronym: TIGER
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 02-274
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2008-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; Pharmacoepidemiology; Quality of Care; Outcomes
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Nearly 2% of veterans >65 are actively treated for epilepsy, and the incidence is projected to increase with the aging of our society. Since commonly used antiepileptic drugs are considered suboptimal for older patients, it is important to understand existing patterns of treatment for older veterans with epilepsy.

DETAILED DESCRIPTION:
OBJECTIVE(S):

1. Identify patient, provider, and system factors predicting adoption of recommended AEDs for treatment of newly diagnosed older veterans (FY00-04).
2. Identify barriers to use of recommended AED in initial therapy for newly diagnosed older veterans with epilepsy.
3. Assess and compare effectiveness of long-term use of various AED.

METHODS:

Using existing national VA outpatient, inpatient, and pharmacy databases in conjunction with Medicare inpatient and outpatient standard analytic files, the 1999 National Health Survey of VA Enrollees, American Hospital Association data, and primary data collection, we will identify the extent to which treatment for older veterans newly diagnosed with epilepsy changed between FY00-FY04, and identify predictors of change at the patient, provider, and system levels. We will begin to identify barriers to use of recommended AED using structured interviews with primary care and general neurology providers in sites with high and low use of suboptimal AEDs in incident cases. Finally, we will compare hospitalizations, emergency room visits, and fall-related injuries (including fractures) for patients on different AED regimens.

RESULTS:

We have identified 72,638 patients who are at least 66 years of age, have a diagnosis of epilepsy in VA or Medicare files, and who also received AEDs from the VA; 9,682 of of these are incident cases, 41,867 are chronic cases, and 21,089 have been defined as having unknown onset. We found wide variations in prescribing, an high rates of use of suboptimal AEDs (70%). We identified sites with high and low use of suboptimal and new AEDs. We have finalized provider interview protocols, and are in the process of gaining approval at individual sites.

IMPACT:

The proposed study will enhance understanding of factors associated with adoption of clinical recommendations for newly diagnosed older patients with epilepsy, begin to identify barriers to their adoption, and assess outcomes of epilepsy patients on chronic AED therapy. This study will provide the foundation on which to develop interventions to improve care and will improve the quality of care for older veterans diagnosed with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

Veterans 66 years and older receiving care from the Veterans Health Administration between fiscal years 2000-2004 Diagnosis of epilepsy and receiving anticonvulsant drugs

Exclusion Criteria:

No VA pharmacy data the year prior to epilepsy diagnosis

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older veterans (66 years and older) with a new diagnosis of epilepsy between 2000-2004
Sampling Method: Non-Probability Sample
Enrollment: 9682 (Actual)
Dates: Start 2000-10; Primary Completion 2004-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Type of Antiepileptic drug prescribed for individuals with new onset epilepsy | Within one year of first epilepsy diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jo Pugh, PhD RN, Principal Investigator — South Texas Health Care System, San Antonio, TX
Locations (2):
- United States (2):
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

REFERENCES:
- [Result] Zeber JE, Copeland LA, Pugh MJ. Variation in antiepileptic drug adherence among older patients with new-onset epilepsy. Ann Pharmacother. 2010 Dec;44(12):1896-904. doi: 10.1345/aph.1P385. Epub 2010 Nov 2. PMID 21045168
- [Result] Pugh MJ, Tabares J, Finley E, Bollinger M, Tortorice K, Vancott AC. Changes in antiepileptic drug choice for older veterans with new-onset epilepsy: 2002 to 2006. J Am Geriatr Soc. 2011 May;59(5):955-6. doi: 10.1111/j.1532-5415.2011.03388.x. No abstract available. PMID 21568976
- [Result] Copeland LA, Ettinger AB, Zeber JE, Gonzalez JM, Pugh MJ. Psychiatric and medical admissions observed among elderly patients with new-onset epilepsy. BMC Health Serv Res. 2011 Apr 19;11:84. doi: 10.1186/1472-6963-11-84. PMID 21504584
- [Result] Pugh MJ, Starner CI, Amuan ME, Berlowitz DR, Horton M, Marcum ZA, Hanlon JT. Exposure to potentially harmful drug-disease interactions in older community-dwelling veterans based on the Healthcare Effectiveness Data and Information Set quality measure: who is at risk? J Am Geriatr Soc. 2011 Sep;59(9):1673-8. doi: 10.1111/j.1532-5415.2011.03524.x. Epub 2011 Aug 10. PMID 21831166
- [Result] Pugh MJ, Berlowitz DR, Rao JK, Shapiro G, Avetisyan R, Hanchate A, Jarrett K, Tabares J, Kazis LE. The quality of care for adults with epilepsy: an initial glimpse using the QUIET measure. BMC Health Serv Res. 2011 Jan 3;11:1. doi: 10.1186/1472-6963-11-1. PMID 21199575
- [Result] Brooks DR, Avetisyan R, Jarrett KM, Hanchate A, Shapiro GD, Pugh MJ, Berlowitz DR, Thurman D, Montouris G, Kazis LE. Validation of self-reported epilepsy for purposes of community surveillance. Epilepsy Behav. 2012 Jan;23(1):57-63. doi: 10.1016/j.yebeh.2011.11.002. Epub 2011 Dec 20. PMID 22189155
- [Result] VanCott AC, Cramer JA, Copeland LA, Zeber JE, Steinman MA, Dersh JJ, Glickman ME, Mortensen EM, Amuan ME, Pugh MJ. Suicide-related behaviors in older patients with new anti-epileptic drug use: data from the VA hospital system. BMC Med. 2010 Jan 11;8:4. doi: 10.1186/1741-7015-8-4. PMID 20064226
- [Result] Ettinger AB, Copeland LA, Zeber JE, Van Cott AC, Pugh MJ. Are psychiatric disorders independent risk factors for new-onset epilepsy in older individuals? Epilepsy Behav. 2010 Jan;17(1):70-4. doi: 10.1016/j.yebeh.2009.10.010. Epub 2009 Nov 12. PMID 19913462
- [Result] Pugh MJ, Vancott AC, Steinman MA, Mortensen EM, Amuan ME, Wang CP, Knoefel JE, Berlowitz DR. Choice of initial antiepileptic drug for older veterans: possible pharmacokinetic drug interactions with existing medications. J Am Geriatr Soc. 2010 Mar;58(3):465-71. doi: 10.1111/j.1532-5415.2010.02732.x. PMID 20398114
- [Result] Pugh MJ, Berlowitz DR, Montouris G, Bokhour B, Cramer JA, Bohm V, Bollinger M, Helmers S, Ettinger A, Meador KJ, Fountain N, Boggs J, Tatum WO 4th, Knoefel J, Harden C, Mattson RH, Kazis L. What constitutes high quality of care for adults with epilepsy? Neurology. 2007 Nov 20;69(21):2020-7. doi: 10.1212/01.WNL.0000291947.29643.9f. Epub 2007 Oct 10. PMID 17928576
- [Result] Berlowitz DR, Pugh MJ. Pharmacoepidemiology in community-dwelling elderly taking antiepileptic drugs. Int Rev Neurobiol. 2007;81:153-63. doi: 10.1016/S0074-7742(06)81009-3. PMID 17433922
- [Result] Pugh MJ, Berlowitz DR, Kazis L. The impact of epilepsy on older veterans. Int Rev Neurobiol. 2007;81:221-33. doi: 10.1016/S0074-7742(06)81014-7. PMID 17433927
- [Result] Zeber JE, Copeland LA, Amuan M, Cramer JA, Pugh MJ. The role of comorbid psychiatric conditions in health status in epilepsy. Epilepsy Behav. 2007 Jun;10(4):539-46. doi: 10.1016/j.yebeh.2007.02.008. Epub 2007 Apr 6. PMID 17416208
- [Result] Pugh MJ, Knoefel JE, Mortensen EM, Amuan ME, Berlowitz DR, Van Cott AC. New-onset epilepsy risk factors in older veterans. J Am Geriatr Soc. 2009 Feb;57(2):237-42. doi: 10.1111/j.1532-5415.2008.02124.x. PMID 19207140
- [Result] Hope OA, Zeber JE, Kressin NR, Bokhour BG, Vancott AC, Cramer JA, Amuan ME, Knoefel JE, Pugh MJ. New-onset geriatric epilepsy care: Race, setting of diagnosis, and choice of antiepileptic drug. Epilepsia. 2009 May;50(5):1085-93. doi: 10.1111/j.1528-1167.2008.01892.x. Epub 2008 Nov 17. PMID 19054416
- [Result] Van Cott AC, Pugh MJ. Epilepsy and the elderly. Annals of Long-Term Care: Clinical Care and Aging. 2008 Jan 1; 16(1):28-32.
- [Result] Pugh MJ, Zeber JE, Copeland LA, Tabares JV, Cramer JA. Psychiatric disease burden profiles among veterans with epilepsy: the association with health services utilization. Psychiatr Serv. 2008 Aug;59(8):925-8. doi: 10.1176/ps.2008.59.8.925. PMID 18678692
- [Result] Pugh MJ, Van Cott AC, Cramer JA, Knoefel JE, Amuan ME, Tabares J, Ramsay RE, Berlowitz DR; Treatment In Geriatric Epilepsy Research (TIGER) team. Trends in antiepileptic drug prescribing for older patients with new-onset epilepsy: 2000-2004. Neurology. 2008 May 27;70(22 Pt 2):2171-8. doi: 10.1212/01.wnl.0000313157.15089.e6. PMID 18505996
- [Result] Pugh MJ, Copeland LA, Zeber JE, Cramer JA, Amuan ME, Cavazos JE, Kazis LE. The impact of epilepsy on health status among younger and older adults. Epilepsia. 2005 Nov;46(11):1820-7. doi: 10.1111/j.1528-1167.2005.00291.x. PMID 16302863
- [Result] Pugh MJ, Foreman PJ, Berlowitz DR. Prescribing antiepileptics for the elderly: differences between guideline recommendations and clinical practice. Drugs Aging. 2006;23(11):861-75. doi: 10.2165/00002512-200623110-00002. PMID 17109565